CLINICAL TRIAL: NCT01040520
Title: Computertomography-based Autopsy (Virtopsy) Versus Conventional Autopsy in Patients Dying in Intensive Care Units
Brief Title: Value of CT-based Autopsy Compared With Conventional Autopsy in ICU Patients
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: UKE KIM 2010.1
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Autopsy
Keywords: CT-based autopsy; virtual autopsy; medical autopsy; quality control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to compare findings generated by CT-based autopsy (Virtopsy) with conventional autopsy and clinical diagnoses. Therefore all patients dying while receiving treatment in the Department of Intensive Care Medicine will be undergo virtopsy and, if relatives give informed consent conventional autopsy.

DETAILED DESCRIPTION:
The aim of the study is to compare findings generated by computertomography-based autopsy (Virtopsy) with conventional autopsy and clinical diagnoses. Therefore all patients dying while receiving treatment in the Department of Intensive Care Medicine will be undergo virtopsy and, if relatives give informed consent conventional autopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients dying in the Department of Intensive Care Medicine while receiving treatment during the study period

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who die while receiving treatment in the Department of Intensive Care Medicine
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

REFERENCES:
- [Derived] Wichmann D, Obbelode F, Vogel H, Hoepker WW, Nierhaus A, Braune S, Sauter G, Pueschel K, Kluge S. Virtual autopsy as an alternative to traditional medical autopsy in the intensive care unit: a prospective cohort study. Ann Intern Med. 2012 Jan 17;156(2):123-30. doi: 10.7326/0003-4819-156-2-201201170-00008. PMID 22250143